CLINICAL TRIAL: NCT05916794
Title: Comparative Effects of Modified Cervical Retraction and Motor Control Therapeutics Exercises on Pain, Range of Motion and Functional Disability in Patients With Cervical Spondylosis
Brief Title: Comparative Effects of Modified Cervical Retraction and Motor Control Therapeutics Exercises in Cervical Spondylosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: : REC/RCR & AHS/23/0123
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Cervical Spondylosis
MeSH Terms: conditions — Spondylosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- : Modified Cervical Retraction Exercises (MCRE) (Experimental): The patient is in sitting OR standing position and faces the physical therapist. The MCRE program consisted of alternating head positions. Hold each position for 20 sec with 8 to 10 repetitions
  Interventions: Other: Modified Cervical Retraction Exercises (MCRE)
- Motor Control therapeutic exercise(MCTE) (Experimental): The MCTE will used is based on retraining the cervical muscles and included four exercises
  Interventions: Other: Motor Control therapeutic exercise(MCTE)

INTERVENTIONS:
Other: Modified Cervical Retraction Exercises (MCRE) — Group A includes Modified cervical retraction exercise The patient is in sitting OR standing position and faces the physical therapist. The MCRE program consisted of alternating head position( neutral, side bending and rotation) while pushing their chin backward patients maintained an upright posture and tried to pull back their shoulders while maintaining this retracted position patient side bend OR rotate their head respectively hold the position for 20 sec.subject performed 5 sets of 10 repetition for 3-4 days per week. Rest intervals of 30 seconds were provided after the completion of 10 repetitions for each pattern and between sets, respectively. The total duration of MCRE will be of approximately 15-20 minutes
  Arms: : Modified Cervical Retraction Exercises (MCRE)
Other: Motor Control therapeutic exercise(MCTE) — Motor control therapeutic exercises will be guided for the retraining of cervical muscles.it include craniocervical flexor exercise,craniocervical extensor exercise, co-contraction of flexors and extensor, a synergy exercise for retraining the strength of the deep neck flexors. Each of these four exercises will be performed for 3 sets of 8 to 10 repetitions, taking an approximate total duration of 15-20 minutes for, 3 days a week
  Arms: Motor Control therapeutic exercise(MCTE)

SUMMARY:
Cervical spondylosis is a general term for age-related wear and tear in the cervical spine that can lead to neck pain, stiffness and other symptoms. Sometimes this condition is called arthritis or osteoarthritis of the neck. The spine likely begins this wearing-down process sometime in your 30s. By age 60, almost nine in 10 people have cervical spondylosis .Objective of this study is to compare the effects of Modified cervical retraction Motor control therapeutic exercises on pain, ROM and functional disability in patients with cervical spondylosis

DETAILED DESCRIPTION:
Cervical spondylosis is a chronic degenerative process of the cervical spine which affects the vertebral bodies and intervertebral discs and causes herniated intervertebral discs, osteophytes, and ligament hypertrophy. It is commonly seen in patients between the ages of 40 and 60. Neck pain not only imposes a notable burden on individuals in the society, but also affects families, the healthcare and economic systems of countries. In 2017, age-standardized prevalence, annual incidence, and years lived with disability from neck pain were estimated at 3551, 807, and 352 per 100,000 population worldwide, respectively Patients seeking medical help for this condition primarily complain of neck pain and/or stiffness. This pain is considered the second most common complaint post low back pain and increased by neck movements especially hyperextension and side bending Currently, there are several therapeutic approaches, either pain relievers or non-medicinal treatments for the management of cervical spondylosis and its associated pain and disability Pain medications mainly include non-steroids anti-inflammatory drugs and narcotics with exercise therapy, massage, physiotherapy, and local injections are among the most common non-medicinal therapies. Evidence suggests that exercise therapy plays a role in improving neck pain and disability of patients with cervical spondylosis. Besides, thanks to being non-invasive and profitable, exercise therapy is commonly used in patient rehabilitation Therapeutic exercises include various workouts such as proprioceptive exercises, stability exercises, strength exercises (dynamic and isometric) and endurance exercises. Neck retraction helps recover the lordotic curve in the lower cervical portion, but kyphotic changes may occur at the upper cervical level. The motor control exercises are the therapeutic approach which mainly focuses on motor control, activation of deep cervical muscles, and aims to retrain the optimal control and coordination of the cervical muscles Apart from the fact that clinical guidelines suggest therapeutic exercises as an integral part of managing neck pain and disability, prescribing the most advantageous exercise therapy has yet been controversial and even current guidelines do not offer specific recommendations on the preferred type and dosage of exercises

ELIGIBILITY:
Inclusion Criteria:

* Age 45 -65 years
* Both. male and female,
* Patient with pain NPRS 4-7
* Subject radiological diagnosed
* Cervical spondylosis (With or without Radiculopathy

Exclusion Criteria:

* Cervical fracture or injury
* Cervical spine osteoporosis,
* Cervical myelopathy & Cervical canal stenosis,
* Cervical Malignancy

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
. Numerical Rating Scale (NPRS) | 6th week
  Numeric Rating Scale (NPRS) is most frequently used instruments to measure pain intensity in neck pain .The 11-point numeric with 0 representing No pain, 1-3 representing Mild Pain (nagging, annoying, interfering little with ADLs), 4-6 representing Moderate Pains (interferes significantly with ADLs), 7-10 representing Sever Pain (disabling, unable to perform ADLs)
Neck Disability Index (NDI) | 6th weeks
  The NDI can be scored as a raw score or doubled and expressed as a percent. Each section is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain. Points summed to a total score The test can be interpreted as a raw score, with a maximum score of 50, or as a percentage.,0 points or 0% means : no activity limitations .50 points or 100% means complete activity limitation. A higher score indicates more patient-rated disability. For patients' understanding, the URDU version is used. A clinically important change was calculated as 5 points, with a sensitivity of 0.78 and a specificity of 0.80
Handheld dynamometry (HHD) | 6th weeks
  A small portable device is held by the examiner and placed against the patient's limb during a maximal isometric contraction. The device can be used to test both proximal and distal muscles in all extremities. Specific dynamometers are used to test grip strength. The Strength measure is more sensitive to change than MMT and correlates well with fixed dynamometry up to 30-kg force. Reliability coefficients for HHD ranged from -0.19 to 0.99, with the majority surpassing 0.70. HHD readings obtained by multiple raters may be up to 53% more variable than those obtained by a single rater

SECONDARY OUTCOMES:
ROM cervical spine (flexion) | 6th weeks
  The patient is seated with upper back supported with chair the center of goniometer is placed over the external auditory meatus, proximal arm is Perpendicular or parallel to ground and distal arm With base of nares or parallel to longitudinal axis of tongue depressor for measuring range of cervical flexion
ROM cervical spine (extension) | 6th weeks
  the center of goniometer is placed over the external auditory meatus, proximal arm is Perpendicular to ground and distal arm With base of nares or parallel to longitudinal axis of tongue depressor and patient extend neck The patient is seated with upper back supported with chair the center of goniometer is placed over the external auditory meatus, proximal arm is Perpendicular or parallel to ground and distal arm With base of nares or parallel to longitudinal axis of tongue depressor and patient extend neck, for measuring the cervical extension ROM.
  [Time Frame: 6th week] The patient is seated with upper back supported with chair the center of goniometer is placed over the external auditory meatus, proximal arm is Perpendicular or parallel to ground and distal arm With base of nares or parallel to longitudinal axis of tongue depressor and pati
ROM cervical spine (side flexion) | 6th weeks
  the center of goniometer is placed Over spinous process of C7,proximal arm over Spinous processes of thoracic vertebrae is perpendicular to ground and distal arm place over Dorsal midline of head. Reference occipital protuberance The patient is seated with upper back supported with chair the center of goniometer is placed Over spinous process of C7,proximal arm over Spinous processes of thoracic vertebrae so that arm is perpendicular to ground and distal arm place over Dorsal midline of head. Reference occipital protuberance for side flexion [Time Frame: 6th week] The patient is seated with upper back supported with chair the center of goniometer is placed Over spinous process of C7,proximal arm over Spinous processes of thoracic vertebrae so that arm is perpendicular to ground and distal arm place over Dorsal midline of head. Reference occipital protuberance for sid
ROM cervical spine (Rotation) | 6th weeks
  the center of the goniometer is placed Over center of cranial aspect of head, proximal arm is placed Parallel to imaginary line between the two acromial processes and distal arm With the tip of the nose. If using the tongue depressor, parallel to the longitudinal axis of tongue depressor for cervical rotation ROM

CONTACTS AND LOCATIONS:
Overall Officials: Sana hafeez, phD*, Principal Investigator — Riphah International University Lahore Campus
Locations (1):
- Riphah Rehabilitation Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lv Y, Tian W, Chen D, Liu Y, Wang L, Duan F. The prevalence and associated factors of symptomatic cervical Spondylosis in Chinese adults: a community-based cross-sectional study. BMC Musculoskelet Disord. 2018 Sep 11;19(1):325. doi: 10.1186/s12891-018-2234-0. PMID 30205836
- [Background] Bernabeu-Sanz A, Molla-Torro JV, Lopez-Celada S, Moreno Lopez P, Fernandez-Jover E. MRI evidence of brain atrophy, white matter damage, and functional adaptive changes in patients with cervical spondylosis and prolonged spinal cord compression. Eur Radiol. 2020 Jan;30(1):357-369. doi: 10.1007/s00330-019-06352-z. Epub 2019 Jul 26. PMID 31350584
- [Background] Rodriguez-Sanz J, Malo-Urries M, Corral-de-Toro J, Lopez-de-Celis C, Lucha-Lopez MO, Tricas-Moreno JM, Lorente AI, Hidalgo-Garcia C. Does the Addition of Manual Therapy Approach to a Cervical Exercise Program Improve Clinical Outcomes for Patients with Chronic Neck Pain in Short- and Mid-Term? A Randomized Controlled Trial. Int J Environ Res Public Health. 2020 Sep 10;17(18):6601. doi: 10.3390/ijerph17186601. PMID 32927858
- [Background] Hidalgo-Perez A, Fernandez-Garcia A, Lopez-de-Uralde-Villanueva I, Gil-Martinez A, Paris-Alemany A, Fernandez-Carnero J, La Touche R. EFFECTIVENESS OF A MOTOR CONTROL THERAPEUTIC EXERCISE PROGRAM COMBINED WITH MOTOR IMAGERY ON THE SENSORIMOTOR FUNCTION OF THE CERVICAL SPINE: A RANDOMIZED CONTROLLED TRIAL. Int J Sports Phys Ther. 2015 Nov;10(6):877-92. PMID 26618067
- [Background] Suni JH, Rinne M, Tokola K, Manttari A, Vasankari T. Effectiveness of a standardised exercise programme for recurrent neck and low back pain: a multicentre, randomised, two-arm, parallel group trial across 34 fitness clubs in Finland. BMJ Open Sport Exerc Med. 2017 Aug 6;3(1):e000233. doi: 10.1136/bmjsem-2017-000233. eCollection 2017. PMID 29021908
- [Background] Lima LV, Abner TSS, Sluka KA. Does exercise increase or decrease pain? Central mechanisms underlying these two phenomena. J Physiol. 2017 Jul 1;595(13):4141-4150. doi: 10.1113/JP273355. Epub 2017 May 26. PMID 28369946
- [Background] Chiarotto A, Maxwell LJ, Ostelo RW, Boers M, Tugwell P, Terwee CB. Measurement Properties of Visual Analogue Scale, Numeric Rating Scale, and Pain Severity Subscale of the Brief Pain Inventory in Patients With Low Back Pain: A Systematic Review. J Pain. 2019 Mar;20(3):245-263. doi: 10.1016/j.jpain.2018.07.009. Epub 2018 Aug 10. PMID 30099210